CLINICAL TRIAL: NCT04965493
Title: A Phase 3 Open-Label, Randomized Study of Fixed Duration Pirtobrutinib (LOXO-305) Plus Venetoclax and Rituximab Versus Venetoclax and Rituximab in Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (BRUIN CLL-322)
Brief Title: A Trial of Pirtobrutinib (LOXO-305) Plus Venetoclax and Rituximab (PVR) Versus Venetoclax and Rituximab (VR) in Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Acronym: BRUIN CLL-322
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18087; J2N-OX-JZNO (Other: Eli Lilly and Company); LOXO-BTK-20022 (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-07-15; First posted 2021-07-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: BTKi; Hematologic Disease; Lymphoma, non-Hodgkin's; Lymphoma, B-cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Diseases; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — pirtobrutinib; venetoclax; Rituximab

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 into Arm A and Arm B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (PVR) (Experimental): Fixed duration pirtobrutinib in combination with venetoclax and rituximab
  Interventions: Drug: Pirtobrutinib; Drug: Venetoclax; Drug: Rituximab
- Arm B (VR) (Active Comparator): Venetoclax with rituximab
  Interventions: Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Pirtobrutinib — Oral
  Other Names: LOXO-305; LY3527727
  Arms: Arm A (PVR)
Drug: Venetoclax — Oral
  Other Names: Venclexta; Venclyxto
Drug: Rituximab — Intravenous (IV)
  Other Names: Rituxan; MabThera; Truxima; Riabni; Ruxience

SUMMARY:
The purpose of this study is to compare the efficacy and safety of fixed duration pirtobruitinib (LOXO-305) with VR (Arm A) compared to VR alone (Arm B) in patients with CLL/SLL who have been previously treated with at least one prior line of therapy. Participation could last up to five years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL/SLL requiring therapy per iwCLL 2018 criteria
* Previous treatment with at least one line of therapy that may include a covalent Bruton's tyrosine kinase (BTK) inhibitor
* Platelets greater than or equal to (≥)50 x 10⁹/liter (L), hemoglobin ≥8 grams/deciliter (g/dL) and absolute neutrophil count ≥1.0 x 10⁹/L
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Estimated creatinine clearance ≥30 milliliters per minute (mL/min)

Exclusion Criteria:

* Known or suspected Richter's transformation at any time preceding enrollment
* Prior therapy with a non-covalent (reversible) BTK inhibitor
* Patients requiring therapeutic anticoagulation with warfarin or another Vitamin K antagonist
* Current treatment with strong cytochrome P450 (CYP) 3A4 (CYP3A4) inhibitors or inducers
* Prior therapy with venetoclax
* Central nervous system (CNS) involvement
* Active uncontrolled systemic bacterial, viral, fungal, or parasitic infection
* Known human immunodeficiency virus (HIV) infection, regardless of cluster of differentiation 4 (CD4) count
* Allogeneic stem cell transplantation (SCT) or chimeric antigen receptor (CAR)-T within 60 days
* Active hepatitis B or hepatitis C
* Known active cytomegalovirus (CMV) infection
* Uncontrolled immune thrombocytopenic purpura (ITP) or autoimmune hemolytic anemia (AIHA)
* Significant cardiovascular disease
* Vaccination with a live vaccine within 28 days prior to randomization
* Patients with the following hypersensitivity:

  * Known hypersensitivity to any component or excipient of pirtobrutinib and venetoclax
  * Prior significant hypersensitivity to rituximab
  * Known allergy to allopurinol and inability to take uric acid lowering agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate progression-free survival (PFS) of pirtobrutinib plus venetoclax and rituximab (Arm A) compared to venetoclax and rituximab (Arm B) | Up to approximately 5 years
  Assessed by blinded independent review committee (IRC) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018

SECONDARY OUTCOMES:
To evaluate the efficacy of Arm A compared to Arm B: Progression-free survival (PFS) | Up to approximately 5 years
  Assessments of efficacy include PFS, assessed by investigator
To evaluate the efficacy of Arm A compared to Arm B: Overall survival (OS) | Up to approximately 5 years
  Assessments of efficacy include OS
To evaluate the efficacy of Arm A compared to Arm B: Time to next treatment (TTNT) | Up to approximately 5 years
  Assessments of efficacy include TTNT
To evaluate the efficacy of Arm A compared to Arm B: Event-free survival (EFS) | Up to approximately 5 years
  Assessments of efficacy include EFS
To evaluate the efficacy of Arm A compared to Arm B: Overall response rate (ORR) | Up to approximately 5 years
  Assessments of efficacy include ORR
To evaluate the efficacy of Arm A compared to Arm B in patient-reported disease-related symptoms | Up to approximately 5 years
  Based on time to worsening of CLL/SLL-related symptoms
To evaluate the efficacy of Arm A compared to Arm B in patient-reported physical functioning | Up to approximately 5 years
  Based on time to worsening of physical functioning

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (176):
- United States (41):
  - Ironwood Physicians, Ironwood Cancer and Research Centers, Chandler, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of California Irvine Medical Center, Orange, California
  - Scripps Mercy Hospital, San Diego, California
  - Providence Medical Foundation, Santa Rosa, California
  - Stamford Hospital, Stamford, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Cancer Specialists of North Florida -St Augustine, Saint Augustine, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - Mission Cancer and Blood, Des Moines, Iowa
  - Pikeville Medical Center, Inc., Pikeville, Kentucky
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Research Medical Center, Kansas City, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - The Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Novant Cancer Institute Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The James Cancer Hospital, Columbus, Ohio
  - Oncology Associates of Bridgeport P.C., Eugene, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - USO - Texas Oncology - San Antonio, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC - Lee Highway, Fairfax, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Swedish Cancer Institute; STE 1020, Seattle, Washington
  - Northwest Cancer Specialists PC, Vancouver, Washington
- Australia (6):
  - Royal Adelaide Hospital, Adelaide
  - Peninsula Private Hospital, Frankston
  - Royal Hobart Hospital, Hobart
  - The Alfred Hospital, Melbourne
  - St Vincent's Hospital, Melbourne
  - Sir Charles Gairdner Hospital, Perth
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Groupe Jolimont, La Louvière
  - CHU UCL Namur site Godinne, Yvoir
- Canada (6):
  - Foothills Medical Centre, Calgary
  - Cross Cancer Institute, Edmonton
  - Jewish General Hospital, Montreal
  - Sunnybrook Research Institute, Toronto
  - BC Cancer Vancouver, Vancouver
  - Cancer Care Manitoba, Winnipeg
- China (27):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Chongqing Cancer Hospital, Chongqing
  - Fujian Provincial Cancer Hospial, Fuzhou
  - Cancer Center of Guangzhou Medical University, Guangzhou
  - First Affiliated Hosp of College of Med, Zhejiang University, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital Of University Of South China, Hengyang
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - The First People's Hospital of Yunnan Province, Kunming
  - Jiangxi Provincial Cancer Hospital, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Nantong Tumor Hospital, Nantong
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai
  - Shanghai Tongren Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - Wu Han Tongji Hospital, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Yichang Central People's Hospital, Yichang
  - Henan Provincial People's Hospital, Zhengzhou
  - Henan Cancer Hospital, Zhengzhou
  - Zhongshan City People's Hospital, Zhongshan
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- Rigshospitalet, Copenhagen, Denmark
- France (12):
  - Centre Hospitalier du Mans, Le Mans
  - Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Morvan
  - CHU de Nantes - Hotel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Hopital de la Pitie Salpetriere, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Pole Regionalde Cancérologie(CHU de Poitiers), Politiers
  - Hôpital de Pontchaillou, Rennes
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen, Rouen
  - ICANS_Institut de Cancerologie Strasbourg Europe, Strasbourg
  - CHRU De Tours, Tours
- Germany (7):
  - Klinikum Chemnitz GmbH, Chemnitz
  - Universtitätsklinikum Essen AöR, Essen
  - Uniklinik Köln, Kerpener
  - München Klinik Schwabing, Koelner Platz 1
  - Universitätsklinikum Leipzig AöR Klinik und Poliklinik für Hämatologie, Leipzig
  - Unimedizin RostockZIM III -Haemtologie, Rostock
  - Gemeinschaftspraxis Dres. Schöttker & Pretscher, z.Hd. Sophie Enz, Würzburg
- Hungary (2):
  - National Institute of Oncology, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Ireland (2):
  - Mater Misericordiae Hospital, Dublin
  - University Hospital Waterford, Waterford
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - IRCCS - AOU di Bologna, Bologna
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - AOU Arcispedale Sant'Anna, Cona
  - Ospedale Santa Croce e Carle, Cuneo
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda Comitato Etico Milano Area C, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - A.O.U. di Modena, Modena
  - Azienda Ospedale Maggiore Della Carita, Novara
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - Policlinico Umberto I - Haematology, Rome
  - A.O.U. Citta' della Salute e della Scienza di Torino, Torino
- Japan (10):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - National Cancer Center Hospital East, Chiba-Ken
  - University of Yamanashi Hospital, Chūō
  - National Cancer Center Hospital, Chūōku
  - University of Fukui Hospital, Fukui
  - Japanese Foundation for Cancer Research, Kōtō City
  - Kyoto Furitsu Medical University Hospital, Kyoto
  - Kochi Medical School Hospital, Nankoku
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
- Norway (2):
  - Akershus Universitetssykehus, Nordbyhagen
  - St-Olavs Hospital, Trondheim
- Poland (7):
  - Szpitale Pomorskie Sp. z o. o., Gdynia
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii, Lodz
  - Klinika Hematoonkologii i Transplantacji Szpiku,Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - MICS Centrum Medyczne Torun, Torun
  - Instytut Hermatologii I Transfuzjologii, Warsaw
- Singapore General Hospital, Singapore, Singapore
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (14):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Puerta De Hierro, Majadahonda
  - Hospital Costa Del Sol, Marbella
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario de Toledo, Toledo
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Skanes Universitetssjukhus, Hematoloaimottagningen, Lund
  - Karolinska Universitetssjukhuset i Solna, Stockholm
- Switzerland (2):
  - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Luzerner Kantonsspital, Lucerne
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (6):
  - Birmingham Heartlands Hospital, Birmingham
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal Marsden Hospital, London
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Trial of Pirtobrutinib (LOXO-305) Plus Venetoclax and Rituximab (PVR) Versus Venetoclax and Rituximab (VR) in Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) (BRUIN CLL-322) — https://trials.lilly.com/en-US/trial/295939